CLINICAL TRIAL: NCT00861939
Title: A Relative Bioavailability Study of Bupropion HCI 300 mg Extended-Release Tablets Under Fasting Conditions
Brief Title: To Demonstrate the Relative Bioavailability of Bupropion HCI 300 mg Extended-Release Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B032032
Record Dates: First submitted 2009-03-12; First posted 2009-03-16 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Bupropion; halofantrine

ARMS (2):
- 1 (Experimental): Bupropion HCl 300mg Extended Release Tablet
  Interventions: Drug: Bupropion HCI 300 mg Extended-Release Tablets EON
- 2 (Active Comparator): WELLBUTRIN XL 300mg Tablets
  Interventions: Drug: WELLBUTRIN XL 300 mg Extended-Release Tablets GlaxoSmithKline

INTERVENTIONS:
Drug: Bupropion HCI 300 mg Extended-Release Tablets EON
  Arms: 1
Drug: WELLBUTRIN XL 300 mg Extended-Release Tablets GlaxoSmithKline
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the relative bioequivalence of Bupropion HCI 300 mg ER Tablets under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B orc.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2004-03; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence according to US FDA timelines | 17 days

CONTACTS AND LOCATIONS:
Overall Officials: So R Hong, M.D., Principal Investigator — Novum Pharmaceutical Research Services